CLINICAL TRIAL: NCT00406393
Title: A Phase III Randomized, Multicenter Trial Comparing Sirolimus/Tacrolimus With Tacrolimus/Methotrexate as Graft-versus-Host Disease (GVHD) Prophylaxis After HLA-Matched, Related Peripheral Blood Stem Cell Transplantation (BMT CTN #0402)
Brief Title: Sirolimus/Tacrolimus Versus Tacrolimus/Methotrexate for Preventing Graft-Versus-Host Disease (GVHD) (BMT CTN 0402)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0402; U01HL069294 (NIH); BMT CTN 0402 (Other: Blood and Marrow Transplant Clinical Trials Network); U01HL069294-05 (NIH)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Leukemia, Myelocytic, Acute; Leukemia, Lymphocytic, Acute; Leukemia, Myeloid, Chronic; Myelodysplastic Syndromes
Keywords: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — Tacrolimus; Methotrexate; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus/Methotrexate (Active Comparator): Patients will be given Tacrolimus and Methotrexate for GVHD prophylaxis.
  Interventions: Drug: Tacrolimus; Drug: Methotrexate
- Tacrolimus/Sirolimus (Experimental): Patients will be given Tacrolimus and Sirolimus for GVHD prophylaxis.
  Interventions: Drug: Tacrolimus; Drug: Sirolimus

INTERVENTIONS:
Drug: Tacrolimus — Adults and Children: Tacrolimus will be given at a dose of 0.02 mg/kg every 24 hours as a continuous intravenous infusion beginning on Day -3. An effort will be made to convert the tacrolimus to oral dosing at 2-3 times the total 24-hour intravenous dose, split into 2 doses given every 12 hours as soon as clinically feasible.
  The target serum level for tacrolimus is 5-10 ng/mL.
  Other Names: Prograf®; FK506
Drug: Methotrexate — Methotrexate will be given at a dose of 15 mg/m2 on Day 1 after transplantation, and at a dose of 10 mg/m2 on Days 3, 6 and 11 after transplantation.
  Other Names: MTX
  Arms: Tacrolimus/Methotrexate
Drug: Sirolimus — Adults: Sirolimus will be given in a loading dose of 12 mg on Day -3 followed by a daily oral dose of 4 mg per day. Doses may be repeated if the subject vomits within 15 minutes of an oral dose.
  Children: Children aged < 12.0 years OR weighing < 40.0 kg will be given an oral loading dose of sirolimus of 3 mg/m2 followed by a daily oral dose of 1 mg/m2, rounded to the nearest full milligram.
  The target serum level for sirolimus is 3-12 ng/mL.
  Other Names: Rapamycin; Rapamune
  Arms: Tacrolimus/Sirolimus

SUMMARY:
The study is designed as a phase III, randomized, open label, multicenter, prospective, comparative trial of sirolimus and tacrolimus versus tacrolimus and methotrexate as graft-versus-host disease (GVHD) prophylaxis after human leukocyte antigen (HLA)-matched, related, peripheral blood stem cell transplantation in individuals with hematologic cancer. Participants will be stratified by transplant center and will be randomly assigned to the sirolimus/tacrolimus or tacrolimus/methotrexate arms at a 1:1 ratio.

DETAILED DESCRIPTION:
BACKGROUND:

Stem cell transplantation is a standard therapy for acute and chronic leukemias and myelodysplastic disorders. A common problem that may occur after a stem cell transplant is a condition known as GVHD. The purpose of this study is to compare two combinations of medications to see which is better at preventing GVHD. The combinations of medications in this study are:

* Sirolimus and tacrolimus
* Methotrexate and tacrolimus

Doctors want to know if one combination is better than the other or if they both have the same result.

DESIGN NARRATIVE:

Participants will receive one of the two conditioning regimens described in the protocol, at the discretion of the transplant physician. The transplant physician must choose among these regimens prior to the participant's assignment to the GVHD prophylaxis treatment. Conditioning regimens will vary by center, but will be the same for all participants at each center. Stem cell donors will donate peripheral blood stem cells according to local institutional practices. Peripheral blood stem cells will not be manipulated or T-depleted prior to administration. Standard post-transplant care will be administered. Participants will be randomly assigned to one of two GVHD prophylaxis regimens and will be followed for the endpoints of interest.

Participants will be followed for 114 days post-randomization for evaluation of the primary endpoint, with additional follow-up for 2 years after transplantation for evaluation of secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 6/6 HLA-matched sibling, defined by Class I (HLA-A and B) serologic typing (or higher resolution) and Class II (HLA-DRBI) molecular typing, who is willing to donate peripheral blood stem cells, and meets institutional criteria for stem cell donation. The donor must be medically eligible to donate stem cells, according to individual transplant center criteria. Pediatric patients for whom a pediatric sibling donor is not anticipated to be a suitable leukapheresis candidate are not eligible.
* Karnofsky performance status of at least 70% or Lansky performance status of at least 70% for participants less than 16 years old
* For participants less than 18 years old, willing and able to take oral medications, per the treating physician's recommendations

Exclusion Criteria:

* Prior allogeneic or autologous transplant using any hematopoietic stem cell source
* Seropositive for the human immunodeficiency virus (HIV)
* Uncontrolled bacterial, viral, or fungal infection (currently taking medication and progression of clinical symptoms)
* Pregnant (positive serum human chorionic gonadotropin [β-HCG] test) or breastfeeding within 4 weeks of study entry
* Kidney function: serum creatinine outside the normal range for age, or measured creatinine clearance less than 50 mL/min/1.72m^2 within 4 weeks of study entry
* Liver function: most recent direct bilirubin, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) greater than two times the upper limit of normal within 4 weeks of study entry
* Lung disease: in adults, forced vital capacity (FVC) or forced expiratory volume in one second (FEV1) less than 60% of predicted value (corrected for hemoglobin); in children, overt hypoxemia, as measured by an oxygen saturation of less than 92% within 4 weeks of study entry
* Cardiac ejection fraction of less than 45% in adults and children, or less than 26% shortening fraction in children within 4 weeks of study entry
* Cholesterol level greater than 500 mg/dL or triglyceride level greater than 500 mg/dL while being treated, or not on appropriate lipid-lowering therapy within 4 weeks of study entry
* Prior history of allergy to sirolimus
* Requires voriconazole at time of study entry
* Currently receiving another investigational drug unless cleared by the protocol officer or protocol chair
* Participants with a history of cancer, other than resected basal cell carcinoma or treated carcinoma in-situ. Cancer treated with curative intent for more than 5 years previously will be allowed. Cancer treated with curative intent for less than 5 years previously will not be allowed unless approved by the protocol officer or protocol chair.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2006-11; Primary Completion 2012-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (24):
- United States (23):
  - City of Hope National Medical Center, Duarte, California
  - UCSD Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - DFCI/Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State, Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University/MCV Hospital, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Hopital Saint-Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.

REFERENCES:
- [Result] Cutler C, Logan B, Nakamura R, Johnston L, Choi S, Porter D, Hogan WJ, Pasquini M, MacMillan ML, Hsu JW, Waller EK, Grupp S, McCarthy P, Wu J, Hu ZH, Carter SL, Horowitz MM, Antin JH. Tacrolimus/sirolimus vs tacrolimus/methotrexate as GVHD prophylaxis after matched, related donor allogeneic HCT. Blood. 2014 Aug 21;124(8):1372-7. doi: 10.1182/blood-2014-04-567164. Epub 2014 Jun 30. PMID 24982504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 2006 to 2011 from 24 different transplant centers.
Period: Overall Study
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Started | 151 | 153
Completed | 149 | 152
Not Completed | 2 | 1
Not completed — Did not undergo transplantation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 59] | 43 [13 to 58] | 44 [13 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 68 | 142
  Male | 77 | 85 | 162
Primary Disease [Number; unit: participants]
  Acute Myelogenous Leukemia (AML) | 71 | 63 | 134
  Acute Lymphoblastic Leukemia (ALL) | 51 | 68 | 119
  Chronic Myelogenous Leukemia (CML) | 9 | 14 | 23
  Myelodysplastic Syndrome (MDS) | 19 | 7 | 26
  Acute Biphenotypic Leukemia (ABL) | 1 | 1 | 2
Disease Status at Transplantation [Number; unit: participants]
  AML 1st Complete Remission | 60 | 56 | 116
  AML 2nd Complete Remission | 11 | 7 | 18
  ALL 1st Complete Remission | 41 | 55 | 96
  ALL 2nd Complete Remission | 10 | 13 | 23
  CML 1st Complete Remission | 7 | 10 | 17
  CML 2nd Complete Remission | 2 | 4 | 6
  ABL 1st Complete Remission | 1 | 1 | 2
  MDS | 19 | 7 | 26
Karnofsky Score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    Scores 90 - 100 | 101 | 116 | 217
    Scores < 90 | 50 | 37 | 87
Recipient-Donor Cytomegalovirus Status [Number; unit: participants] — Seropositivity (+) or Seronegativity (-) for the recipient / Seropositivity (+) or Seronegativity (-) for the donor
  participants
    +/+ | 59 | 47 | 106
    +/- | 14 | 24 | 38
    -/+ | 30 | 44 | 74
    -/- | 38 | 30 | 68
    Missing | 10 | 8 | 18
Conditioning Regimen [Number; unit: participants]
  Cyclophosphamide/Total Body Irradiation | 124 | 122 | 246
  Etoposide/Total Body Irradiation | 27 | 31 | 58

OUTCOME MEASURES:

1. Primary Outcome: Rate of Grades II-IV Acute GVHD-free Survival
Description: The primary objective is to compare rates of 114-day Grades II-IV acute GVHD-free survival post randomization for HLA-matched, related donor allogeneic peripheral blood stem cell transplantation using two different GVHD prophylaxis regimens. Participants are graded on a scale of 1 to 4 according to their symptoms and organs involved, where 4 represents a worse grade.
Time Frame: Day 114
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 67 [59 to 74] | 62 [54 to 70]

2. Secondary Outcome: Incidence of Acute GVHD
Description: Cumulative incidence of acute GVHD (grade II-IV) occurring 100 days from transplantation.
Time Frame: Measured at Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 26 [19 to 34] | 34 [26 to 41]

3. Secondary Outcome: Time to Neutrophil and Platelet Engraftment
Description: Neutrophil engraftment is defined as achieving an Absolute Neutrophil Count (ANC) > 500/mcL for three consecutive measurements on different days. Platelet engraftment is defined as a platelet count > 20,000/mcL for three consecutive measurements over three or more days.
Time Frame: Measured through Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
days
  Neutrophil Engraftment | 14 [8 to 27] | 16 [10 to 68]
  Platelet Engraftment | 16 [7 to 100] | 19 [9 to 100]

4. Secondary Outcome: Mucositis Severity
Description: Mucositis severity will be scored per the modified Oral Mucositis Assessment Scale (OMAS) scoring system on a scale of 0 - 4, where 0 equals normal mucosa and 4 represents severe mucosa.
Time Frame: Measured at Day 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
units on a scale | 0.31 (0.28) | 0.47 (0.40)

5. Secondary Outcome: Rate of Veno-occlusive Disease (VOD)
Description: VOD will be defined as the occurrence of VOD (based on the Baltimore Criteria for the diagnosis of VOD) in conjunction with other end-organ dysfunction.
Time Frame: Measured through Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 11 [6 to 16] | 5 [2 to 9]

6. Secondary Outcome: Thrombotic Microangiopathy (TMA) Infection
Description: The occurrence of TMA within the first 100 days after stem cell transplantation will be recorded. The first day of onset will be used for reporting purposes.
Time Frame: Measured through Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 5 [3 to 10] | 1 [0 to 4]

7. Secondary Outcome: Reactivation of Cytomegalovirus (CMV) Infection
Time Frame: Measured at Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 13 [9 to 19] | 15 [10 to 21]

8. Secondary Outcome: Treatment-related Mortality
Time Frame: Measured at Day 100 and Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants
  Day 100 | 7 [3 to 11] | 7 [4 to 12]
  Year 2 | 20 [13 to 26] | 16 [11 to 23]

9. Secondary Outcome: Malignant Disease Relapse
Description: Testing for recurrent malignancy in the blood, marrow or other sites will be used to assess relapse after transplantation. For the purpose of this study, relapse is defined by either morphological or cytogenetic evidence of AML, ALL, CML, MDS or CMML consistent with pre-transplant features.
Time Frame: Measured at Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 28 [20 to 35] | 29 [22 to 37]

10. Secondary Outcome: Overall Survival
Time Frame: Measured at Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 149 | 152
percentage of participants | 59 [51 to 67] | 63 [55 to 70]

11. Secondary Outcome: Infections
Time Frame: Measured at Year 2
Population: Insufficient data to report on this outcome measure
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Time to Discharge After Transplant
Time Frame: Measured at Year 2
Population: Insufficient data to report on this outcome measure
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2-years post transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event.
Arm/Group | Tacrolimus/Sirolimus | Tacrolimus/Methotrexate
Serious Adverse Events (participants affected / at risk) | 9/149 | 12/152
Other Adverse Events (participants affected / at risk) | 0/149 | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus/Sirolimus (N=149) | Tacrolimus/Methotrexate (N=152)
Mental status changes (Psychiatric disorders) | 1 (1) | 0
Death (General disorders) | 1 (1) | 0
Embolism (Vascular disorders) | 1 (1) | 0
Aphasia (Nervous system disorders) | 1 (1) | 0
Thoracotomy (Surgical and medical procedures) | 1 (1) | 0
Retinal tear (Eye disorders) | 1 (1) | 0
Chest pain (General disorders) | 1 (1) | 0
Staphylococcal infection (Infections and infestations) | 1 (1) | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 (1)
Septic shock (Infections and infestations) | 0 | 1 (1)
Glaucoma (Eye disorders) | 0 | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-12-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT00406393/Prot_SAP_ICF_000.pdf